CLINICAL TRIAL: NCT04892719
Title: 4DX Functional Lung Imaging in the Diagnosis of Chronic Lung Allograft Dysfunction After Lung Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: 4DMedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00103179
Record Dates: First submitted 2021-04-29; First posted 2021-05-19 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Lung Transplant; Complications
Keywords: Lung Transplantation; Chronic Lung Allograft Dysfunction

STUDY DESIGN:
Intervention Model Description: This study uses a case control design and approximately 15 lung transplant recipients will be enrolled (10 CLAD cases/5 CLAD free controls). The study procedures will be performed during a single research visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Participants who underwent a lung transplant at Duke (Other): Participants will undergo fluoroscopic chest imaging with 4Dx technology software analysis
  Interventions: Diagnostic Test: Fluoroscopic chest imaging with 4Dx technology software analysis

INTERVENTIONS:
Diagnostic Test: Fluoroscopic chest imaging with 4Dx technology software analysis — 4DxV utilizes a novel software algorithm to analyze data from cinefluoroscopy images to calculate regional ventilation and pulmonary function changes. Cinefluorography uses a fluorescent screen with X-rays to make real-time moving images the lung described below. This is the same x-ray fluoroscopy that is used in clinical imaging and the fluoroscopic imaging time is approximately 1 minute leading to an effective radiation dose of 2 mSv (200 mRem). This is significantly lower that the radiation exposure from a standard chest CT. Fluoroscopy images are acquired at each of five views for approximately enough time to capture at least one complete, continuous breath. The subject is required to remain in the same position for each of the five fluoroscopy imaging sequences. These images will be analyzed by the novel 4Dx technology to provide the 4Dx lung function analysis report.

SUMMARY:
This is a pilot study to determine the utility of Novel Functional Lung Imaging and Ventilation (4DxV) Analysis software in measurement of lung ventilation abnormalities and diagnosis of chronic lung allograft dysfunction (CLAD) after lung transplantation.

DETAILED DESCRIPTION:
This is a pilot study to determine the feasibility and utility of Novel Functional Lung Imaging and Ventilation (4DxV) Analysis software in measurement of lung ventilation abnormalities and diagnosis of CLAD after lung transplantation. 4DxV is a technology developed by 4Dx (4Dx Limited, Melbourne, Australia and Los Angeles, CA) and is a novel computational approach to the data obtained from standard fluoroscopic imaging that measures tissue motion of the lung at all locations and in all phases of breath. These motion measurements are used to calculate 4-dimensional ventilation (4DxV) of lung tissue to provide variety of outputs. The investigators will establish the sensitivity, specificity, and accuracy of this technology in diagnosis of CLAD compared to CT scan and pulmonary function results in patients with a known diagnosis of CLAD based on established diagnostic criteria.

The investigators will test the following hypotheses:

1. 4DxV scans will be able to detect quantitative ventilation abnormalities in patients with established CLAD and the severity of the abnormalities will correlate with severity of PFT decline
2. 4DxV will be able to diagnose patients with CLAD of the bronchiolitis obliterans syndrome (BOS) phenotype grades 0 (CLAD free) vs grades 1-3

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years of age at the time of written informed consent
2. Recipient of a first bilateral lung transplantation performed at Duke University at least one year prior to written informed consent
3. Computed tomography (CT) scan of the chest performed at Duke as standard of care after transplantation but within 1 year prior to written informed consent 4a. CLAD grades 1, 2,or 3 (per ISHLT 2014 criteria [Meyer et al 2014]) prior to or at the time of screening

   * Grade 1 is defined as a fractional decrease in FEV1 to 66-80% of post-transplant baseline FEV1
   * Grade 2 is defined as a fractional decrease in FEV1 to 51%-65% of post-transplant baseline FEV1
   * Grade 3 is defined as a fractional decrease in FEV1 to <= 50% of post-transplant baseline FEV14b. CLAD free status (defined as most recent FEV1 at the time of screening >90% of post-transplant baseline FEV1)

Exclusion Criteria:

1. Recipients of a single lung transplant
2. Recipients of a redo-lung transplant
3. Recipients of bone marrow or stem cell transplant
4. Recipients of a multi-organ transplant
5. Patients with hospital admissions(excluding admissions for planned treatment of the CLAD and/or rejection)within one month of screening.
6. Patients who are unable to lie flat on the fluoroscopy table
7. Pregnant women (by subject's verbal report). Lung transplant recipients are routinely counseled to avoid pregnancy due to the teratogenic effects of necessary immunosuppressant medications. Pregnancy after lung transplantation is therefore extremely rare. As this is a minimal risk study which does not involve an experimental therapy, invasive devices, or increased risk procedures, pregnancy testing is deemed unnecessary for this population for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Ventilation defect percentage (VDP) as measured by XV lung ventilation analysis software | At least one year after lung transplantation
  Determine the VDP using XV Lung Ventilation Analysis Software to quantify ventilation in lung transplant patients
Regional ventilation heterogeneity percentage as measured by XV lung ventilation analysis software | At least one year after lung transplantation
  Determine the ventilation heterogeneity percentage using XV Lung Ventilation Analysis Software to quantify ventilation in lung transplant patients

SECONDARY OUTCOMES:
Calculation of Bronchiolitis Obliterans Syndrome (BOS) Stage based on FEV1 decline | At least one year after lung transplantation
  Determine BOS stage based on subject's pulmonary function test measurements of percent FEV1 decline compared to post transplant baseline FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Azfar Ali, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meyer KC, Raghu G, Verleden GM, Corris PA, Aurora P, Wilson KC, Brozek J, Glanville AR; ISHLT/ATS/ERS BOS Task Force Committee; ISHLT/ATS/ERS BOS Task Force Committee. An international ISHLT/ATS/ERS clinical practice guideline: diagnosis and management of bronchiolitis obliterans syndrome. Eur Respir J. 2014 Dec;44(6):1479-503. doi: 10.1183/09031936.00107514. Epub 2014 Oct 30. PMID 25359357